CLINICAL TRIAL: NCT05231720
Title: Mannheim Register of Sepsis and Septic Shock
Acronym: MARSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Michael Behnes, Prof. Dr., Universitätsmedizin Mannheim
Other Study IDs: 2019-694N
Record Dates: First submitted 2021-01-13; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Severe Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to investigate clinically and prognostically relevant parameters in patients with sepsis and septic shock within a monocentric observational clinical register.

DETAILED DESCRIPTION:
All consecutive septic patients at the internists intensive care Unit (ICU) at the University of Mannheim are included in the register and follow up during ICU stay and after that. Data of patients' admission status, septic focus, baseline parameters, and comorbidities are collected. Extensive information about echocardiography, electrocardiography, and imaging procedures are included in the register. Laboratory values, microbiological investigations, organ dysfunction and organ replacement therapies, medication, adverse events, and complications were recorded for several days during the ICU stay (days 1, 2,3, 5,7, and 10). Standard scores for critically ill patients were calculated for the day before admission at the ICU if available, and several time points during the ICU stay. The register includes information about the mortality during ICU stay, 30-day mortality, 6-month mortality, and septic patients' 1-year mortality.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis and septic shock according to current guidelines

Exclusion Criteria:

* other forms of shock not associated with an infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes internal medicine patients presenting sepsis and septic shock at the ICU irrespective of the septic focus.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-12-03 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | 30 days

SECONDARY OUTCOMES:
all-cause mortality | in hospital
all-cause mortality | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Medical Centre Mannheim, Mannheim, Baden-Wurttemberg
  - First Department of Medicine, University Medical Centre Mannheim, Mannheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Forner J, Weidner K, Rusnak J, Dudda J, Behnes M, Akin I, Schupp T. Prognostic Impact of Left Compared to Right Heart Function in Sepsis and Septic Shock. ASAIO J. 2024 Jun 1;70(6):502-509. doi: 10.1097/MAT.0000000000002131. Epub 2024 Jan 18. PMID 38237636